CLINICAL TRIAL: NCT00540345
Title: Four Arms, Multicenter, Open Label Study of Tailored Regimens With Peginterferon Plus Ribavirin for Genotype 2 Chronic Hepatitis C
Brief Title: Four Arms, Multicenter Study of Tailored Regimens With Peginterferon Plus Ribavirin for Genotype 2 Chronic Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, MING-LUNG,YU, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUH-IRB-960057
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Hepatitis C
Keywords: chronic hepatitis C; genotype 2; rapid virological response; sustained virological response; peginterferon; ribavirin; treatment duration
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A, RVR LD RBV (Active Comparator): Patients who have a RVR will be randomized into two groups with a ratio of 1:1 (Arm A & B)B, RVR SD RBV A, RVR LD RBV B, RVR SD RBV
  Interventions: Drug: pegylated interferon alpha 2a and plus ribavirin
- B, RVR SD RBV (Active Comparator): Patients who have a RVR will be randomized into two groups with a ratio of 1:1 (Arm A & B)B, RVR SD RBV
  Interventions: Drug: Pegylated interferon alfa-2a and ribavirin
- C, non-RVR 24w (Active Comparator): For patients who do not have a RVR will be randomized into two groups with a ratio of 1:1 (Arm C & D) (C, non-RVR 24w) (D, non-RVR 48w)
  Interventions: Drug: pegylated interferon alpha 2a and ribavirin
- D, non-RVR 48w (Active Comparator): For patients who do not have a RVR will be randomized into two groups with a ratio of 1:1 (Arm C & D)(C, non-RVR 24w) (D, non-RVR 48w)
  Interventions: Drug: pegylated interferon alpha 2a and ribavirin

INTERVENTIONS:
Drug: pegylated interferon alpha 2a and plus ribavirin — pegylated interferon alpha 2a 180 mcg/week and Ribavirin 1000-1200 mg/day for 4 weeks followed by pegylated interferon alpha 2a 180 mcg/week and Ribavirin 800 mg/day for 12 weeks, follow up for 24 weeks
  Other Names: PEGASYS®
  Arms: A, RVR LD RBV
Drug: Pegylated interferon alfa-2a and ribavirin — pegylated interferon alfa-2a 180 mcg/week and Ribavirin 1000-1200 mg/day for 16 weeks, follow up for 24 weeks
  Other Names: PEGASYS®
  Arms: B, RVR SD RBV
Drug: pegylated interferon alpha 2a and ribavirin — pegylated interferon alpha 2a 180 mcg/week and Ribavirin 1000-1200 mg/day for 24 weeks, follow up for 24 weeks
  Other Names: PEGASYS®
  Arms: C, non-RVR 24w
Drug: pegylated interferon alpha 2a and ribavirin — pegylated interferon alpha 2a 180 mcg/week and Ribavirin 1000-1200 mg/day for 48 weeks, follow up for 24 weeks
  Other Names: PEGASYS®
  Arms: D, non-RVR 48w

SUMMARY:
The purposes of this study are:

1. To evaluate the efficacy and safety of low-dose versus standard-dose of ribavirin in combination with peginterferon alfa-2a given for 16 weeks in hepatitis C virus (HCV) genotype 2 infected, treatment-naïve chronic hepatitis C patients after achieving a rapid virologic response (RVR,defined as seronegativity of HCV RNA at week 4 of treatment).
2. To evaluate the efficacy and safety of 24-week versus 48-week regimen of peginterferon alfa-2a plus standard-dose of ribavirin in HCV genotype 2 infected, treatment-naïve chronic hepatitis C patients who have no RVR.

DETAILED DESCRIPTION:
The recommended regimen for treating HCV genotype 2 patients is peginterferon plus low dose ribavirin (800 mg/day) for 24 weeks. Recently studies have demonstrated that a shorter treatment duration of 12-16 weeks of peginterferon plus standard weight-based dose of ribavirin (800-1400 mg/day) is as effective as a 24-week regimen among HCV genotype 2 patients with a RVR at week 4 of treatment (rate of sustained virological response, SVR, approximately 90%). However, for patients without a RVR at week 4 the efficacy of 24 week treatment remains unsatisfied. Individualized therapy with tailored regimen according to baseline and on-treatment virological factors, without compromising efficacy, is the future strategy in the management of chronic hepatitis C.

The aims of the present study are

1. To evaluate the efficacy and safety of low-dose versus standard-dose of ribavirin in combination with peginterferon alfa-2a given for 16 weeks in hepatitis C virus (HCV) genotype 2 infected, treatment-naïve chronic hepatitis C patients after achieving a rapid virologic response (RVR,defined as seronegativity of HCV RNA at week 4 of treatment).
2. To evaluate the efficacy and safety of 24-week versus 48-week regimen of peginterferon alfa-2a plus standard-dose of ribavirin in HCV genotype 2 infected, treatment-naïve chronic hepatitis C patients who have no RVR.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years of age
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribavirin
* Serologic evidence of chronic hepatitis C infection by an anti-HCV antibody test
* Detectable serum HCV-RNA and HCV viral genotype 2
* Liver biopsy findings consistent with the diagnosis of chronic hepatitis C infection with or without compensated cirrhosis (Exception: hemophiliacs in whom biopsy is medically contra-indicated do not require biopsy.)
* Compensated liver disease (Child-Pugh Grade A clinical classification)
* Negative urine or blood pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of study drug
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment and during the 6 months after treatment end

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding
* Therapy with any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug
* Any investigational drug 6 weeks prior to the first dose of study drug
* Co-infection with active hepatitis A, hepatitis B and/or human immunodeficiency virus (HIV)
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* Signs or symptoms of hepatocellular carcinoma
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count < 1500 cells/mm3 or platelet count < 90,000 cells/mm3 at screening
* Serum creatinine level > 1.5 times the upper limit of normal at screening
* History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration)
* Evidence of drug abuse (including excessive alcohol consumption) within one year of study entry
* Inability or unwillingness to provide informed consent or abide by the requirements of the study
* Male partners of women who are pregnant
* Hgb < 11 g/dL in women or < 12 g/dL in men at screening
* Any patient with major thalassemia
* Patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled if, in the judgment of the investigator, an acute decrease in hemoglobin by up to 4 g/dL (as may be seen with ribavirin therapy) would not be well-tolerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2006-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Efficacy - Rapid virologic response (RVR), HCV RNA seronegative by PCR at week 4 Sustained virological response (SVR), HCV RNA seronegative by PCR throughout 24-week off-treatment period | 1.5 year

SECONDARY OUTCOMES:
Safety - adverse event rate and profile | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Lung Yu, MD, PhD, Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Mangia A, Santoro R, Minerva N, Ricci GL, Carretta V, Persico M, Vinelli F, Scotto G, Bacca D, Annese M, Romano M, Zechini F, Sogari F, Spirito F, Andriulli A. Peginterferon alfa-2b and ribavirin for 12 vs. 24 weeks in HCV genotype 2 or 3. N Engl J Med. 2005 Jun 23;352(25):2609-17. doi: 10.1056/NEJMoa042608. PMID 15972867
- [Background] Dalgard O, Bjoro K, Hellum KB, Myrvang B, Ritland S, Skaug K, Raknerud N, Bell H. Treatment with pegylated interferon and ribavarin in HCV infection with genotype 2 or 3 for 14 weeks: a pilot study. Hepatology. 2004 Dec;40(6):1260-5. doi: 10.1002/hep.20467. PMID 15558712
- [Background] von Wagner M, Huber M, Berg T, Hinrichsen H, Rasenack J, Heintges T, Bergk A, Bernsmeier C, Haussinger D, Herrmann E, Zeuzem S. Peginterferon-alpha-2a (40KD) and ribavirin for 16 or 24 weeks in patients with genotype 2 or 3 chronic hepatitis C. Gastroenterology. 2005 Aug;129(2):522-7. doi: 10.1016/j.gastro.2005.05.008. PMID 16083709
- [Background] Yu ML, Dai CY, Huang JF, Hou NJ, Lee LP, Hsieh MY, Chiu CF, Lin ZY, Chen SC, Hsieh MY, Wang LY, Chang WY, Chuang WL. A randomised study of peginterferon and ribavirin for 16 versus 24 weeks in patients with genotype 2 chronic hepatitis C. Gut. 2007 Apr;56(4):553-9. doi: 10.1136/gut.2006.102558. Epub 2006 Sep 6. PMID 16956917
- [Background] Strader DB, Wright T, Thomas DL, Seeff LB; American Association for the Study of Liver Diseases. Diagnosis, management, and treatment of hepatitis C. Hepatology. 2004 Apr;39(4):1147-71. doi: 10.1002/hep.20119. No abstract available. PMID 15057920